CLINICAL TRIAL: NCT00558532
Title: Omega-3 Fatty Acid Status in Morbid Obesity Before and After Surgical Treatment
Status: Withdrawn | Type: Observational
Why Stopped: Investigator Retired.
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, J. Wesley Alexander, Emeritus, University of Cincinnati
Other Study IDs: 07-66
Record Dates: First submitted 2007-11-14; First posted 2007-11-15 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Morbid Obesity; Cardiovascular Disease; Fatty Acid Levels
Keywords: Morbid obesity; Omega-3 fatty acid levels
MeSH Terms: conditions — Obesity, Morbid; Cardiovascular Diseases | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, fat tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Surgical: Those subjects undergoing bariatric surgery or abdominal surgery following a previous bariatric surgery.
  Interventions: Procedure: Bariatric Surgery
- Control: Volunteers who have dietary habits similar to the subjects.

INTERVENTIONS:
Procedure: Bariatric Surgery — Open roux-en-Y gastric bypass, open banded sleeve gastrectomy, abdominoplasty, other abdominal surgery
  Groups: Surgical

SUMMARY:
The purpose of this study is to determine the concentration of omega-3 fatty acids in plasma, blood and abdominal fat before and after bariatric surgery to provide guidance for future studies.

DETAILED DESCRIPTION:
The omega-3 fatty acids are essential for human growth, development and well-being. Numerous studies have shown that a relatively high intake of the omega-3 fatty acids are beneficial in brain and visual development, psychiatric disorders, rheumatic disorders, inflammatory responses and cardiovascular disease. As an example, low levels of tissue omega-3 fatty acids are associated with a markedly higher rate of death from cardiac causes compared to patients with relatively high concentrations of the omega-3 fatty acids. Obese patients often have an unhealthy dietary intake and evidence of increased inflammatory processes. After a gastric bypass patients will have decreased absorption of fats from the gastrointestinal tract and may become fatty acid deficient. While gastric bypass may decrease death from cardiovascular disease in morbidly obese patients, cardiovascular disease is still the most common cause of death after a gastric bypass. There are numerous nutritional deficiencies which occur after gastric bypass and many of these are well documented. However, there are no data concerning the plasma and tissue levels of omega-3 fatty acids in morbidly obese patients either before or after operation.

ELIGIBILITY:
Inclusion Criteria:

* Surgical group candidates must be undergoing surgery for morbid obesity, abdominoplasty or other abdominal operation.
* Must have adequate venous access.

Exclusion Criteria:

* Insufficient venous access

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing an operation for morbid obesity will be candidates for inclusion in the study as will all candidates who are undergoing abdominoplasty or other abdominal operations post bariatric surgery.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Omega-3 Fatty acid levels in whole blood, plasma and abdominal fat sample | Within 3 months of surgery

CONTACTS AND LOCATIONS:
Overall Officials: J. W. Alexander, M.D., Principal Investigator — UC Surgeons Center fo Surgical Weight Loss/ University of Cincinnati
Locations (1):
- The Christ Hospital, Cincinnati, Ohio, United States